CLINICAL TRIAL: NCT06422039
Title: A Clinical Study to Evaluate the Relative Bioavailability of HRS-7535 Tablets of Different Formulating Processes and the Effects of Food on New Formulates (Single Center, Random, Open, Cross)
Brief Title: Bioavailability and Food Effects of HRS-7535 Tablets With Different Formulating Processes in Healthy Subjects
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shandong Suncadia Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HRS-7535-103
Record Dates: First submitted 2024-05-14; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study was an open, fixed-sequence clinical trial in healthy adult subjects
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment group A (Experimental)
  Interventions: Drug: HRS-7535（D）Tablets; Drug: HRS-7535（C）Tablets
- Treatment group B (Experimental)
  Interventions: Drug: HRS-7535（D）Tablets; Drug: HRS-7535（C）Tablets
- Treatment group C (Experimental)
  Interventions: Drug: HRS-7535（D）Tablets; Drug: HRS-7535（C）Tablets

INTERVENTIONS:
Drug: HRS-7535（D）Tablets — One HRS-7535（D）Tablet is administered to healthy subjects.
Drug: HRS-7535（C）Tablets — Two HRS-7535（C）Tablets is administered to healthy subjects.

SUMMARY:
This study was designed as a a single-center, randomized, open, interleaved (3-cycle, 3-sequence) trial. It is planned to enroll 18 healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent;
2. Male or female aged 18-45 at screening (both inclusive);
3. Male weight ≥ 50 kg, female weight ≥ 45 kg, and body mass index (BMI) : 18-30 kg/m2 (including both ends of the value);
4. Subjects (including male subjects) are willing to have no birth plan and voluntarily adopt effective contraceptive measures and no sperm donation plan from Signed informed consent to the last two weeks after the administration of no fertility plan and no sperm donation, egg donation plan, and agree to take effective contraceptive measures.

Exclusion Criteria:

1. Those who had a smoking history in the 3 months before screening (average daily smoking > 5 cigarettes), or could not stop using any tobacco products during the test;
2. Those who consumed an average of more than 25 g of alcohol per day (e.g., 750 mL beer, 250 mL wine, or 50 mL liquor) in the three months prior to screening, or who could not abstain during the trial period;
3. Consumed any beverage or food containing grapefruit in the 7 days prior to screening; Or consumed any beverage or food containing methylxanthine within 2 days prior to screening, such as coffee, tea, cola, chocolate, etc.
4. Allergy, or suspected allergy to any ingredient in HRS-7535 preparation;
5. A history of drug abuse in the past five years or use of drugs in the three months prior to the test; Or a positive urine drug test;
6. A history of any clinically serious disease or disease or condition that the investigator believes may affect the test results, including but not limited to circulatory, endocrine, nervous, digestive, urinary, or blood, immune, psychiatric, or metabolic disorders;
7. Abnormalities with QTcF > 450 ms detected by 12-lead electrocardiogram at screening or baseline and judged by investigators to be clinically significant;
8. Vital signs, physical examination, laboratory examination, abdominal ultrasound or chest imaging examination at the time of screening or at baseline suggest abnormalities that the investigators have determined to be clinically significant;
9. Positive hepatitis B surface antigen (HBsAg), positive antibodies against hepatitis C virus (HCV), positive antibodies against human immunodeficiency virus (HIV), or positive antibodies against syphilis within 4 weeks prior to screening;
10. Use of any prescription, over-the-counter, herbal or dietary supplements (excluding regular vitamins) in the 2 weeks prior to screening;
11. Participants in clinical trials of any other drug or medical device within the 3 months prior to screening or within the 5 half-life of the drug (based on whether the drug was administered or used, excluding placebo);
12. Received BCG vaccine within 12 months prior to screening; Vaccination or exposure to other live or attenuated vaccines (other than COVID-19 vaccines) within 3 months prior to screening; Or who plan to be vaccinated during the trial;
13. Patients who have had any surgery in the 3 months prior to screening, have not recovered from surgery, or are likely to have surgery or hospitalization plans during the trial period;
14. Blood donation (or blood loss) and blood donation (or blood loss) ≥400 mL within 3 months before screening, or receiving blood transfusion;
15. Positive results of serum pregnancy test (serum beta-HCG test) during screening period or baseline examination in women;
16. The woman had any form of pregnancy (including spontaneous abortion, delivery, ectopic pregnancy, etc.) in the 3 months prior to the screening, or was breastfeeding at the time of the screening visit;
17. Women use the following contraceptive methods during screening visits: medicated extended-release Iuds, extended-release contraceptives (subcutaneous implants, vaginal rings, microspheres and microcapsules); Use of long-acting contraceptive injections before screening (medroxyprogesterone acetate should be prohibited 3 months before screening, other injections should be prohibited 1 month before screening), use of oral contraceptives 2 months before screening, and use of contraceptive patches 1 month before screening; Special cases are judged by the researcher;
18. Subjects have conditions that, as determined by the investigator, affect drug absorption, distribution, metabolism, and excretion, or reduce adherence, or other factors that make participation in the study inappropriate.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
PK parameters：Cmax | 0 hour to 72 hours after the last dosing
PK parameters：AUC0-t | 0 hour to 72 hours after the last dosing
PK parameters：AUC0-∞ | 0 hour to 72 hours after the last dosing
Relative bioavailability of HRS-7535 (D) tablets compared to HRS-7535 (C) tablets following a high-fat meal | 0 hour to 72 hours after the last dosing
Relative bioavailability of HRS-7535 (D) tablets under both fasting and fed (high fat meal) status | 0 hour to 72 hours after the last dosing

SECONDARY OUTCOMES:
PK parameters：Tmax | 0 hour to 72 hours after the last dosing
PK parameters： t1/2 | 0 hour to 72 hours after the last dosing
PK parameters： CL/F | 0 hour to 72 hours after the last dosing
PK parameters： V/F | 0 hour to 72 hours after the last dosing
Incidence and severity of adverse events (AEs) | from screening to 72 hours after the last dosing

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical Uniersity, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided